CLINICAL TRIAL: NCT06074445
Title: An Anonymous Survey Investigating Care for the Sexual Health of Cancer Survivors and Their Intimate Partners, as Provided by the United Kingdom Hospital Cancer Team
Brief Title: Caring for the Sexual Health and Wellbeing of Cancer Survivors and Their Intimate Partners: An Anonymous Survey
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: National Institute for Health Research, Applied Research Collaboration, Wessex (Unknown); Fortuneswell Cancer Trust (Unknown); Dorset County Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: Ethics ID 39453
Record Dates: First submitted 2023-08-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Cancer
Keywords: Cancer Survivors; Neoplasms; Oncology; Sexual Health; Sexual Dysfunction, physiological; Sexual Dysfunctions, psychological; Sexuality; Barrier; Facilitator; Professional-Patient Relations; Communication
MeSH Terms: conditions — Neoplasms; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Sexuality; Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with Cancer: No intervention
  Interventions: Other: No intervention
- Partners of People with Cancer: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this survey study is to provide broad information as reported by cancer survivors and their intimate partners about both their sexual health and their experiences of care from the United Kingdom hospital cancer team, including their perspectives on factors that may hinder or help care. This information will be analysed and used to inform the questions asked in a separate, subsequent, qualitative study.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer survivors diagnosed with any type of cancer at age 18 years or over
2. A partner of someone diagnosed with any type of cancer at age 18 years or over
3. Cancer diagnosis must be no more than 10 years ago
4. Cancer survivors or their partners who experienced treatment and follow up care in the United Kingdom

Exclusion Criteria:

1. Cancer survivors who were diagnosed with cancer below the age of 18 years
2. Partners of cancer survivors who were diagnosed with cancer below the age of 18 years
3. Cancer diagnosis was more than 10 years ago
4. Cancer survivors/partners of survivors where the cancer treatment and follow up was not in the United Kingdom
5. Previous completion of the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with cancer or the partners of people with cancer
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who had a sexual health discussion(s) with the hospital cancer team at any point during cancer care | Up to 10 years prior to completing survey (discussion(s) about sexual health could have occurred at any point during cancer care)
  Sexual health discussion:19 examples of the sort of topics that may have been discussed in relation to sexual health

SECONDARY OUTCOMES:
Number of participants with specific levels of impact on their sex lives by cancer and its treatments | From each individual participants' cancer diagnosis/cancer treatment until the date that they completed the survey
  As above
Survey questionnaire to measure the nature and prevalence of care for sexual health that cancer survivors and their intimate partners self-report experiencing from the UK hospital cancer team. | Participants can report care received from prior to their cancer treatment through to their follow-up care (last 10 years only)
  An online survey questionnaire (no validated questionnaire available and therefore research created the questionnaire based on a literature reviews on sexual health in oncology
Survey questionnaire to measure the nature and prevalence of the perceived barriers to and facilitators for care for sexual health as received by cancer survivors and their intimate partners when provided by the UK hospital cancer team. | Participants can report their perceptions from diagnosis through to their follow-up care (last 10 years only)
  As above
Survey questionnaire to measure to what extent groups of cancer survivors and their intimate partners with differing characteristics receive differing care for their sexual health from the UK hospital cancer team. | Participants diagnosed with cancer in the previous 10 years.
  Participants' responses from outcomes 1-4 will be used toinform this outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sam Porter, PhD, RN, Principal Investigator — Bournemouth University
Locations (1):
- Bournemouth University, Bournemouth, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant information sheet stated that information would not be made publicly available via a data sharing repository. This approach was taken due to the sensitive nature of the topic and was anticipated to provide reassurance and potentially improve recruitment.

REFERENCES:
- [Derived] Sheppard S, Culliford D, Glen T, Lee S, Sheppard ZA, Porter S. Care for sexual health in oncology survey: a regression analysis of variables associated with the likelihood of people with cancer having a sexual health discussion with the hospital cancer team. Eur J Oncol Nurs. 2025 Oct;78:102977. doi: 10.1016/j.ejon.2025.102977. Epub 2025 Sep 1. PMID 40967121